CLINICAL TRIAL: NCT05035966
Title: Association of Plasma β-amyloid 40 and 42 With Risk of Prediabetes
Brief Title: Association of β-amyloid 40 and 42 With Prediabetes
Status: Completed | Type: Observational
Sponsor: Liegang Liu (Other)
Responsible Party: Sponsor-Investigator, Liegang Liu, Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: XBP20210903
Record Dates: First submitted 2021-09-03; First posted 2021-09-05 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: PreDiabetes
Keywords: β-amyloid 40; β-amyloid 42; prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prediabetes: In the case-control study, prediabetes was diagnosed according to the diagnostic criteria recommended by the WHO in 1999. Prediabetes was defined as impaired fasting glucose (FPG ≥6.1 mmol/L and <7.0 mmol/L, and 2-h post-glucose load <7.8 mmol/L) and/or impaired glucose tolerance (FPG <6.1 mmol/L, and 2-h post-glucose load ≥7.8 mmol/L and <11.1 mmol/L). In the nested case-control study, new-onset prediabetes was defined as FPG ≥6.1 mmol/L and <7.0 mmol/L.
  Interventions: Other: Plasma β-amyloid 40 and 42 concentration
- Healthy control: In the case-control study, healthy control was defined as FPG <6.1 mmol/L and 2-h post-glucose load <7.8 mmol/L. In the nested case-control study, healthy control was defined as FPG <6.1 mmol/L.
  Interventions: Other: Plasma β-amyloid 40 and 42 concentration

INTERVENTIONS:
Other: Plasma β-amyloid 40 and 42 concentration — Plasma β-amyloid 40 and 42 concentrations were simultaneously measured by validated assay platforms from Meso Scale Discovery (MSD; Rockville, MD, USA).

SUMMARY:
Background: Previous epidemiological and animal studies have suggested a strong relationship between prediabetes and Alzheimer's disease. Recently, we demonstrated that plasma β-amyloid (Aβ), a potential biomarker for Alzheimer's disease, was elevated in individuals with type 2 diabetes. However, few studies have investigated the associations of plasma Aβ40 and Aβ42 concentrations with prediabetes.

Objective: we aimed to investigate the associations of plasma Aβ40 and Aβ42 concentrations with risk of prediabetes in two independent studies.

Design: We performed a case-control study and a nested case-control study within a prospective cohort study. In the case-control study, we included 571 newly diagnosed individuals with prediabetes and 571 control participants. Prediabetes individuals were consecutively recruited from subjects who attended the outpatient clinics of Department of Endocrinology at Tongji Medical College Hospital from 2012 to 2015. Concomitantly, we recruited healthy controls from a general population undergoing a routine health checkup in the same hospital. One healthy control was selected at random for each prediabetes individuals according to age (±3 years) and sex. The inclusion criteria of participants were as follows: age ≥30 and ≤80 years, BMI <40 kg/m2, no history of prediabetes and diabetes mellitus, no history of receiving pharmacological treatment for hyperlipidemia, nor any clinically systemic disease, any acute illness, and chronic inflammatory or any infective disease. An independent nested case-control study was conducted within an ongoing cohort study, namely the Tongji-Ezhou cohort. Briefly, 5533 participants, including 3101 retired employees and 2432 working employees, were enrolled from Echeng Stell and received healthcare for a baseline investigation between 2013 and 2015. The first follow-up for all participants was finished by mid-2020. Considering the low incidence of prediabetes among young working employees, we performed the nested case-control study among retired employees. During the follow-up, 119 new-onset prediabetes cases were diagnosed within the retired employees according to fasting plasma glucose. We randomly selected the control participants who matched 2:1 to the cases by age (±3 years) and sex from the retired employees with normal fasting plasma glucose. The inclusion criteria were the same as the case-control study; 2 new-onset prediabetes cases aged >80 years were excluded. Additionally, 17 cases without enough plasma were excluded. Finally, 100 individuals with new-onset prediabetes and 200 well-matched control participants were included for the analysis of the nested case-control study. These two studies were approved by the Ethics and Human Subject Committee of Tongji Medical College. All enrolled participants in the two studies were of Chinese Han ethnicity and provided informed written consent. Plasma Aβ40 and Aβ42 concentrations were simultaneously measured by validated assay platforms from Meso Scale Discovery (MSD; Rockville, MD, USA).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥30 and ≤80 years, BMI <40 kg/m2, screened for prediabetes or diabetes, and with enough plasma collected for β-amyloid 40 and 42 detection.

Exclusion Criteria:

* History of diabetes mellitus and prediabetes, pharmacological treatment for hyperlipidaemia, any clinically systemic disease, any acute illness, chronic inflammatory disease or any infective disease.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the participants enrolled were of Chinese Han ethnicity. They gave informed written consent to the study and did not take any medication known to affect glucose tolerance or insulin secretion before participation.
Sampling Method: Probability Sample
Enrollment: 1442 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Prediabetes | Newly diagnosed prediabetes in the case-control study was diagnosed between 2012 and 2015; new-onset prediabetes in the nested case-control study was identified between 2013 and 2020.
  In the case-control study, prediabetes was diagnosed in accordance with the diagnostic criteria recommended by WHO in 1999; in the nested case-control study, new-onset prediabetes was confirmed as FPG ≥7.0 mmol/l.